CLINICAL TRIAL: NCT03117374
Title: The Impact of an Innovative Web-based School Nutrition Intervention to Increase Fruits and Vegetables and Dairy Products in Adolescents
Brief Title: Impact of Web-based School Nutrition Intervention to Increase Fruits, Vegetables and Dairy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laval University (Other)
Responsible Party: Principal Investigator, Vicky Drapeau, Associate Professor, Laval University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: FO096053
Record Dates: First submitted 2017-04-04; First posted 2017-04-17 (Actual); Last update posted 2017-04-17 (Actual); Status verified 2017-04

CONDITIONS: Eating Behavior
MeSH Terms: conditions — Feeding Behavior

STUDY DESIGN:
Who Masked: Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Team Nutriathlon intervention (Experimental): Participants were invited to participate in the Team Nutriathlon for an 8-week period
  Interventions: Behavioral: Team Nutriathlon intervention
- Control (No Intervention): Participants were invited to follow the regular school curricular for an 8-week period

INTERVENTIONS:
Behavioral: Team Nutriathlon intervention — 8 wk web-based nutrition intervention program aimed at increasing the consumption of fruits, vegetables and dairy products.
  Arms: Team Nutriathlon intervention

SUMMARY:
The goal of this study is to evaluate the impact of an innovative web-based school nutrition intervention (Team Nutriathlon) aimed at promoting the consumption of vegetables and fruit and dairy products in high school students and to identify facilitators and/or barriers influencing its success.

DETAILED DESCRIPTION:
Classes of first and second year secondary students (grades 9 and 10) from the Québec City region will be randomized into two groups. Participants in the intervention (Team Nutriathlon) will be asked to increase their consumption of fruits and vegetables and dairy products using an innovative web-based platform, developed for this study, over six weeks. The control group will follow the regular school curriculum. The number of servings of fruits and vegetables and dairy products consumed by students per day and facilitators and barriers influencing the success of the program will be compared between the two groups over the study.

ELIGIBILITY:
Inclusion Criteria:

* Schools were recruited on a voluntary basis via email invitation and sent across the region of Québec. The selected schools were of medium to high socioeconomic levels according to the Deprivation Index of the Ministry of Education of Québec.

Exclusion Criteria:

* None

Ages: 13 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 282 (Actual)
Dates: Start 2011-09-09 (Actual); Primary Completion 2013-06-23 (Actual); Study Completion 2013-08-30 (Actual)

PRIMARY OUTCOMES:
Change in fruits and vegetables and dairy products | Before and after the intervention (0 and 6 wk)
  Change in the servings of fruits and vegetables and milk and alternatives assessed with a web-based questionnaire

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chamberland K, Sanchez M, Panahi S, Provencher V, Gagnon J, Drapeau V. The impact of an innovative web-based school nutrition intervention to increase fruits and vegetables and milk and alternatives in adolescents: a clustered randomized trial. Int J Behav Nutr Phys Act. 2017 Oct 16;14(1):140. doi: 10.1186/s12966-017-0595-7. PMID 29037203